CLINICAL TRIAL: NCT07072260
Title: Investigation of the Effect of Activator-Assisted Talocrural Joint Manipulation on Acute Sports Performance Parameters in Elite Male Volleyball Players
Brief Title: Effect of Activator-Assisted Talocrural Manipulation on Performance in Elite Volleyball Players
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara Yildirim Beyazıt University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2025/047
Record Dates: First submitted 2025-07-09; First posted 2025-07-18 (Actual); Last update posted 2025-07-18 (Actual); Status verified 2025-07

CONDITIONS: Joint Manipulation; Range of Motion; Athletic Performance; Sports; Balance; Jumping Performance; Physical Therapy Modalities; Postural Balance; Motor Activity; Volleyball
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Single Blind (Statistician analyzing data was blinded)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Activator-Assisted Talocrural Manipulation (Experimental): Participants in this group receive a single session of activator-assisted manipulation using the Activator Adjustment Instrument (AAI) to the talocrural (ankle) joint. Six impulses (three anterior and three posterior) are applied with the ankle in a neutral position.
  Interventions: Other: Activator Manipulation
- Sham Soft Tissue Stroking (Sham Comparator): Participants in this group receive a sham intervention consisting of light soft tissue stroking around the talocrural joint without joint manipulation. The application mimics the duration and setup of the experimental group but does not include any mechanical stimulus.
  Interventions: Other: Sham Stroking

INTERVENTIONS:
Other: Sham Stroking — Participants in this group receive a sham intervention consisting of light soft tissue stroking around the talocrural joint without joint manipulation. The application mimics the duration and setup of the experimental group but does not include any mechanical stimulus.
  Other Names: Non-therapeutic light touch technique
  Arms: Sham Soft Tissue Stroking
Other: Activator Manipulation — Participants in this group receive a single session of activator-assisted manipulation using the Activator Adjustment Instrument (AAI) to the talocrural (ankle) joint. Six impulses (three anterior and three posterior) are applied with the ankle in a neutral position.
  Other Names: Activator Adjustment Instrument (AAI)
  Arms: Activator-Assisted Talocrural Manipulation

SUMMARY:
This randomized controlled trial aims to evaluate the acute effects of activator-assisted talocrural joint manipulation on joint range of motion, dynamic balance, vertical and horizontal jump performance, and weight transfer parameters in elite male volleyball players aged 18-25. The study compares a manipulation group with a sham control group and assesses performance metrics before and after the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Elite male volleyball players aged 15-25 years
* Minimum of 3 years of professional volleyball training experience
* Active member of a team and club

Exclusion Criteria:

* Not actively participating in training or matches
* History of acute musculoskeletal pathology or surgery in the lower extremities

Ages: 15 Years to 25 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes — Elite male volleyball players aged 15-25 years
Enrollment: 60 (Actual)
Dates: Start 2025-05-10 (Actual); Primary Completion 2025-05-20 (Actual); Study Completion 2025-05-30 (Actual)

PRIMARY OUTCOMES:
Ankle Range of Motion (Plantar/Dorsiflexion) | Pre-intervention (T0) and post-intervention (T1, within 3-5 minutes).
  Plantar and dorsiflexion measured using a goniometer (degrees).
Y-Balance Test | Pre-intervention (T0) and post-intervention (T1, within 3-5 minutes).
  Anterior, posteromedial, and posterolateral reach distances (cm).
Jumping Performance: | Pre-intervention (T0) and post-intervention (T1, within 3-5 minutes).
  Vertical jump height and horizontal jump distance (cm).
Dynamic Weight Transfer | Pre-intervention (T0) and post-intervention (T1, within 3-5 minutes).
  Assessed via pedobarographic analysis, including static load ratio (%), dynamic contact area ratio (CAR-AP, CAR-RP, %), and dynamic speed (mm/s).

CONTACTS AND LOCATIONS:
Locations (1):
- Gazi University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared due to privacy concerns and institutional data protection policies.

REFERENCES:
- [Derived] Haksever B, Hajighorbani K, Cakir CH, Isguzar MG, Elbasan B. Investigation of the effect of activator-assisted talocrural joint manipulation on acute sports performance parameters in elite male volleyball players. BMC Sports Sci Med Rehabil. 2025 Oct 7;17(1):291. doi: 10.1186/s13102-025-01358-1. PMID 41053891